CLINICAL TRIAL: NCT05726110
Title: A Single-arm Open-label Multicenter Clinical Study of Selinexor in Combination With HAD or CAG Rregimens in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Selinexor in Combination With HAD or CAG Rregimens in Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Collaborators: Antengene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanxiBethuneH
Record Dates: First submitted 2023-01-29; First posted 2023-02-13 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — selinexor; Homoharringtonine; Daunorubicin; Cytarabine; Granulocyte Colony-Stimulating Factor; aclacinomycins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selinexor、HAD or CAG regimens (Experimental): * Selinexor (60 mg) is used twice weekly for two weeks (four times, 240 mg total of selinexor) in combination with HAD or CAG regimens for reinduction therapy in patients with relapsed and refractory AML.
  * (Bone marrow image indicates active hyperplasia) HAD regimen: homoharringtonine (HHT) (2mg/ m^2/d)×7days, daunorubicin (DNR, 40mg/ m^2/d)×3 days, cytarabine (Ara-C,100-200mg/ m^2/d)×7 days (no leukocyte drugs should be used throughout the treatment process)；
  * (Bone marrow image indicates hypoproliferation)CAG regimen: Granulocyte Colony-Stimulating Factor (G-CSF, 5ug/kg/d, started 12 hours before chemotherapy×14 days (d1-d14), aclacinomycin (20mg/d)×4 days (d1-4), cytarabine (10 mg/ m^2, subcutaneous injection, 1 time in 12 hours)×14 days (d1-d14).
  * G-CSF was discontinued in the CAG regimen when WBC > 20×10^9/L, but chemotherapy was not stopped.
  Interventions: Drug: Selinexor; Drug: Homoharringtonine; Drug: Daunorubicin; Drug: Cytarabine; Drug: Granulocyte Colony-Stimulating Factor; Drug: Aclacinomycin

INTERVENTIONS:
Drug: Selinexor — Given PO
  Other Names: KPT-330
Drug: Homoharringtonine — Given per standard of care
  Other Names: HHT
Drug: Daunorubicin — Given per standard of care
  Other Names: DNR
Drug: Cytarabine — Given per standard of care
  Other Names: Ara-C
Drug: Granulocyte Colony-Stimulating Factor — Given per standard of care
  Other Names: G-CSF
Drug: Aclacinomycin — Given per standard of care
  Other Names: ACM

SUMMARY:
This clinical trial studies the efficacy and safety of selinexor combined with HAD or CAG regimen in the treatment of relapsed or refractory acute myeloid leukemia

DETAILED DESCRIPTION:
Main Purpose：

To observe the efficacy of selinexor in combination with HAD or CAG regimen for relapsed and refractory acute myeloid leukemia :complete remission rate (CR rate), partial remission rate (PR rate), no remission rate (NR rate), complete remission with incomplete hematologic recovery(CRi rate)

Secondary Purposes：

1. To observe the recurrence rate of selinexor combined with HAD or CAG regimen for relapsed and refractory acute myeloid leukemia, treatment-related mortality(TRM), Overall Survival (OS), Event-Free Survival (EFS);
2. Safety indicators: to observe adverse events and deaths during treatment with selinexor in combination with HAD or CAG regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-60 years old;
2. Except for patients with AML-M3 with acute myeloid leukemia；
3. Meet the diagnostic criteria for refractory AML (2011 Chinese guidelines for the diagnosis and treatment of acute myeloid leukemia (relapsed or refractory)):(1) The standard regimen did not achieve complete remission after 2 courses of induction chemotherapy;(2) Relapse within 6 months after the first complete remission; (3) Patients who relapse after 6 months after the first complete remission, and those who fail to induce chemotherapy after the original program; (4) 2 or more recurrences; (5) Extramedullary leukemia persists；
4. Meet the diagnostic criteria for recurrent AML (refer to the 2014 NCCN guidelines): after complete remission, (1) naive cells appear in peripheral blood; (2) >5% of bone marrow naive cells; (3) Extramedullary recurrence；
5. The bone marrow image indicates active hyperplasia or hypoproliferation；
6. Eastern Oncology Collaborative Group Physical Status Assessment (ECOG-PS) with a score of 0-2.

Exclusion Criteria:

1. Accompanied by cerebral hemorrhage；
2. Pregnancy；
3. Have a mental illness or other condition that cannot proceed as planned；
4. Severe arrhythmia, abnormal ECG (QT>500ms).

Early withdrawal from test criteria：

Participants have the right to withdraw from the study at any time from the trial. Exit Criteria:

1. The subject or the subject's legally authorized representative requests to withdraw from the study;
2. Participant loss to follow-up.

Doctor/Investigator required subjects to terminate the trial early:

1. Subjects who are unable to carry out follow-up treatment due to adverse events (serious irreversible organ function damage during treatment) who are judged by the investigator to be unsuitable for continuing the research;
2. The subject does not adhere to the protocol, such as the use of chemotherapy drugs, etc., which affects the effectiveness and safety judgment.

For participants who withdrew early from the study (except subjects who were lost to follow-up), the reason for their early withdrawal should be recorded, and the time of the last study's medication/treatment should be recorded, and the examination items at the time of early withdrawal from the study should be completed at the last visit, if possible.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-29 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission Rate | max 2 years
  complete remission rate(CR rate), partial remission rate (PR rate) , no remission rate (NR rate)

SECONDARY OUTCOMES:
Recurrence Rate | max 2 years
  After complete remission, (1) naive cells appear in peripheral blood; (2) >5% of bone marrow naive cells; (3) Extramedullary recurrence(refer to the 2014 NCCN guidelines).
Treatment-Related Mortality (TRM) | max 2 years
  A death that is considered to be causally linked to a treatment
Overall Survival (OS) | max 2 years
  Overall survival is a secondary endpoint that will be measured as time from the start of treatment until death from any cause, or the last date the patient was known to be alive
Event-Free Survival (EFS) | max 2 years
  Event-free survival (EFS) was calculated from the time of informed consent until death, not achieving CR/CRi or relapse after CR/CRi.
Safety:Incidence and severity of adverse events | max 2 years
  To evaluate the possible adverse events and deaths during treatment with selinexor in combination with HAD or CAG，mainly including liver toxicity, cardiotoxicity, bacterial infection, viral infection, fungal infection.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, Study Director — Shanxi Bethune Hospital Regulatory Authority
Locations (1):
- Tao Wang, Taiyuan, Shanxi, China

DOCUMENTS (1):
  • Study Protocol (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT05726110/Prot_000.pdf